CLINICAL TRIAL: NCT04918472
Title: Minimally Invasive Evaluation of Dyspepsia by Combined Magnetically Controlled Capsule Endoscopy and Urea Breath Test: a Pilot Prospective Cohort Study
Acronym: MCUDYSPEPSIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Assitant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021.194
Record Dates: First submitted 2021-06-03; First posted 2021-06-08 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Dyspepsia; Peptic Ulcer Disease; Gastroesophageal Reflux; Ugi Malignancies; Pancreatobiliary Disease
MeSH Terms: conditions — Dyspepsia; Peptic Ulcer; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCCE (Experimental): Magnetically controlled capsule endoscopy will be performed before UGI endoscopy.
  Interventions: Procedure: MCCE

INTERVENTIONS:
Procedure: MCCE — Mangetically controlled capsule endoscopy will be performed

SUMMARY:
The combined diagnostic accuracy of MCCE and UBT in Hong Kong patients with uninvestigated dyspepsia between age 35 to 60 years for structural pathology and HP infection is comparable to that of conventional UGI endoscopy with histological examination for HP

DETAILED DESCRIPTION:
Dyspepsia affects about 20% of the population globally and represents one of the commonest reasons for patients to seek medical consultation.1-3 The definition of dyspepsia has evolved over time and generally encompasses a variety of upper gastrointestinal (UGI) symptoms that can be of anatomical or functional origin such as epigastric pain or burning, bloating, postprandial fullness, belching, early satiety and nausea.2, 4 While diagnostic criteria (eg, Rome IV criteria) have been proposed to better characterize and standardize symptoms of functional dyspepsia for research purpose, there is considerable overlap of clinical presentation between functional dyspepsia and organic / anatomical causes of dyspeptic symptoms such as peptic ulcer disease (PUD), gastroesophageal reflux disease (GERD), UGI malignancies, or pancreatobiliary diseases.2, 3, 5, 6 Therefore, it is of clinical importance to differentiate clinically significant anatomical pathologies from functional disorders during the initial evaluation of patients with dyspeptic symptoms.

Society guidelines based on Western population data with a relatively lower prevalence of helicobacter pylori (HP) and UGI cancers (eg, cancer of stomach, esophagus) generally recommend an initial noninvasive management approach (eg, "test and treat" strategy for HP and empiric trial of acid suppressive therapy) in dyspeptic patients without alarming symptoms or age < 50 - 60, and reserve upfront endoscopy for high-risk patients with alarming symptoms (eg, gastrointestinal bleeding, iron deficiency anemia, dysphagia, unintended weight loss, etc) or age ≥ 50 - 60.2, 3 However, in Asian populations with a relatively higher prevalence of HP and UGI cancers, an initial noninvasive management approach to dyspeptic symptoms based on alarming symptoms and age cutoff at 50 - 60 years may not be entirely appropriate since up to 25% of patients with UGI cancers may not have alarming symptoms.7 In a recent systematic review with meta-analysis of dyspepsia management in Asian countries, alarming symptoms and age were found to be poor predictors of UGI cancers and 17.8% of dyspeptic patients who were eventually diagnosed with UGI cancers were younger than age 45.6

In a study of 5066 UGI endoscopies performed in Asian patients with dyspepsia, clinically significant structural pathologies (PUD, cancers of stomach / esophagus, esophagitis) were found in 19.5% of patients.8 Although UGI endoscopy is the gold standard for diagnosis of clinically significant structural pathologies and HP infection by histology, it is an invasive procedure with a small but finite risk of complication.3 When compared to the invasive nature of conventional UGI endoscopy, an initial minimally invasive diagnostic approach that can evaluate for both UGI structural pathology and HP infection would be highly desirable and clinically relevant in Asian patients with uninvestigated dyspepsia between 35 to 60 years of age.

Wireless capsule endoscopy (CE) (commonly known to the general public as the "pill camera") represents a minimally invasive diagnostic modality for visualization of the gastrointestinal (GI) tract and is well tolerated by patients.9 While conventional CE has been shown to provide adequate visualization of luminal pathologies in the small bowel, colon and esophagus, visualization of the different parts of stomach by conventional CE remains challenging due to its passive propulsion through the GI tract by peristalsis or gravity and the large cavity size of the stomach. Recently, magnetically controlled capsule endoscopy (MCCE) systems comprised of small capsule endoscope, guidance magnet robot, data recorder, and computer workstation for real-time viewing and control of CE have become available and can provide a more controlled visualization of different anatomical parts of the stomach by CE.10, 11 In a study of 350 patients with UGI symptoms requiring conventional UGI endoscopy for evaluation, MCCE was shown to be safe and was able to provide adequate visualization of the stomach with a high sensitivity (90.4%) and specificity (94.7%) for focal gastric lesions when compared with conventional UGI endoscopy.11 However, despite its promising role as a minimally invasive diagnostic modality for structural pathologies of stomach, MCCE does not allow tissue acquisition and thus cannot provide information on HP infection status by rapid urease test (RUT) or histological examination. On the other hand, noninvasive test for HP by urea breath test (UBT) has been shown to be highly sensitive and specific for HP infection and can supplement MCCE to provide important information on the status of HP infection.12

To date, there has been no dedicated study on the use of combined MCCE and UBT for minimally invasive evaluation of dyspepsia in Asian population. In order to address the gap in knowledge, we would like to propose a pilot prospective cohort study to investigate the clinical utility of combined MCCE and UBT as the initial minimally invasive evaluation of uninvestigated dyspepsia in Hong Kong patients between 35 to 60 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 60
* Patients with uninvestigated dyspeptic symptoms including epigastric pain or burning, bloating, postprandial fullness, belching, early satiety and nausea
* Patients who are able to provide written informed consent to participate in the study and comply with the study procedures.

Exclusion Criteria:

* Unable to provide written informed consent
* Patients with contraindications for conventional UGI endoscopy or MCCE due to comorbidities
* Patients with dysphagia, gastroparesis, gastrointestinal (GI) tract obstruction, or surgically altered anatomy of the GI tract
* Patients with a permanent pacemaker, or implantable cardioverter-defibrillator
* Patients with any electronic/magnetic/mechanically controlled devices e.g. sacral nerve stimulators, bladder stimulators
* Patients with known inflammatory bowel disease, cancer of the GI tract
* Patients who are pregnant or lactating

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The combined diagnostic accuracy of MCCE and UBT as gold standard | 2 weeks
  The combined diagnostic accuracy of MCCE and UBT in Hong Kong patients with uninvestigated dyspepsia between age 35 to 60 years for structural pathology and HP infection using conventional UGI endoscopy and histological examination for HP as gold standard

SECONDARY OUTCOMES:
The sensitivity and specificity of MCCE for clinically significant structural pathology in UGI (defined as peptic ulcers, cancers, reflux esophagitis) as gold standard | during endoscopy
  The sensitivity and specificity of MCCE for clinically significant structural pathology in UGI (defined as peptic ulcers, cancers, reflux esophagitis) in Hong Kong patients with uninvestigated dyspepsia between age 35 to 60 years using conventional UGI endoscopy as gold standard
The sensitivity and specificity of UBT for HP infection in Hong Kong patients with uninvestigated dyspepsia between age 35 to 60 years using histological examination for HP by UGI endoscopy as gold standard | during endoscopy
  The sensitivity and specificity of UBT for HP infection in Hong Kong patients with uninvestigated dyspepsia between age 35 to 60 years using histological examination for HP by UGI endoscopy as gold standard
Adverse events up to 2 weeks after UBT, MCCE, UGI endoscopy | 2 weeks after endoscopy
  Adverse events up to 2 weeks after UBT, MCCE, UGI endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No